CLINICAL TRIAL: NCT02954835
Title: Negative Pressure Therapy for Closed Groin Wounds in Patients Undergoing Vascular Surgery
Brief Title: Negative Pressure Therapy for Groin Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-16-679
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena (Active Comparator): Subjects randomized to the Prevena dressing will have the dressing in place for 5 to 7 days postoperatively and removed before discharge, or at the first outpatient visit.
  Interventions: Device: Prevena
- Traditional Dressing (Active Comparator): Subjects randomized to the traditional dressing will undergo dressing changes as per the standard protocol with the first dressing change at postoperative day 2 or 3, or at the discretion of the attending surgeon.
  Interventions: Device: Traditional Dressing

INTERVENTIONS:
Device: Prevena — Prevena is a sterile silver dressing. On top of the silver dressing is an adhesive plastic, which is connected to a therapy unit through a short length suction tube.
  Arms: Prevena
Device: Traditional Dressing — Sterile gauze dressing secured by tape.
  Arms: Traditional Dressing

SUMMARY:
The purpose of this study is to compare wound infection rates between negative pressure therapy (Prevena) and the traditional sterile dry dressing among patients undergoing vascular surgery involving groin incisions.

DETAILED DESCRIPTION:
This is a prospective, investigator-initiated, post-market data collection study comparing wound infection rates among patients undergoing vascular surgery involving groin incisions. Patients will be randomized on the day of surgery to receive the traditional sterile dry dressing or Prevena. Patients with the traditional dressing will undergo dressing changes as per the standard protocol with the first dressing change at postoperative day 2 or 3, or at the discretion of the attending surgeon. The patients with Prevena dressing will have the dressing in place for 5 to 7 days postoperatively and removed before discharge, or at the first outpatient visit. The Primary Objective of this study is to see if using negative pressure therapy decreases the rate of infection. The Secondary Objectives will include multivariate analysis to understand which patients may have a compounded benefit from Prevena (e.g. smokers, diabetics, and obese patients). The Prevena System is an FDA approved bandage and will be used in this study for on-label purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vascular surgery with a groin incision.

Exclusion Criteria:

* Allergy to silver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12; Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Infection rate | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bernik, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: hospital public website — http://www.englewoodhealth.org